CLINICAL TRIAL: NCT03382327
Title: Multicentric Study Determining the Benefit of the Use of 3D Models and Tools in Hepatectomy Planning for Hepatocarcinomas
Brief Title: Benefit of the Use of 3D Models and Tools in Hepatectomy Planning for Hepatocarcinomas
Acronym: 3D-HAPPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-003
Record Dates: First submitted 2017-11-14; First posted 2017-12-22 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Hepatocarcinoma
Keywords: Surgical planning; CT-scan; MRI; 3D model; Hepatocarcinoma eligible for surgical resection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical planning (Experimental): Two surgical plans will be established preoperatively. The first plan will be based on standard preoperative images (CT-scan, MRI) review. The second plan will be based on the 3D model review.
  Interventions: Procedure: Surgical planning

INTERVENTIONS:
Procedure: Surgical planning — Two surgical plans will be established preoperatively. The first plan will be based on standard preoperative images (CT-scan, MRI) review. The second plan will be based on the 3D model review. Both will be compared to the actual surgery performed in the operating room.

SUMMARY:
The aim of this study is to assess the benefit of 3D models in the planning of hepatic resection by comparing the changes in the surgical plan based on the analysis of conventional preoperative images (CT-scan and MRI), compared to the surgical plan based on the analysis of 3D reconstruction.

DETAILED DESCRIPTION:
The detailed anatomical description of the liver described by Couinaud in 1954 is the basis for hepatic surgery. Surgical resection is the approach leading to the best survival rate in case of liver cancer. In hepatocarcinomas, systematic removal of the infected liver segment is considered the most effective technique to eliminate tumour, potential satellite nodules and avoid vascular spread. Resectability rate highly depends on the analysis of preoperative images. However, in 20% of cases, there are modifications compared with the initial surgical plan leading to an increase in morbidity rate.

In 2002, Couinaud highlighted the difficulty of identifying portal pedicles, especially because of anatomical variations, and recommended the use of a three-dimensional reconstruction from images provided by a helical scanner.

The hypothesis of the study is that 3D models would improve surgical planning leading to a decrease in intra-operative adjustments and mortality.

The aim of this multicentric, prospective study is to assess the benefit of 3D models in the surgical management of hepatocarcinomas, more specifically in the detailed analysis of 3D vascular structures and in the surgery planning with resection merges evaluation. The validation of this virtual method will be built on the comparison of the surgical plan based on the analysis of conventional preoperative images (CT-scan and MRI) and the surgical plan based on the analysis of 3D reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a hepatocarcinoma, eligible for surgical resection
* Patient over 18 years old
* Patient able to understand the study and provide written informed consent
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patient with other liver tumours
* Patient whose general condition is not suitable for study participation (WHO ≥ 3)
* Patient with a condition preventing its participation to study procedures, according to investigator's judgment
* Patient with contraindications to injected CT-scan or MRI: allergic reaction to contrast agents, kidney failure, pacemaker, claustrophobia
* Pregnancy or breastfeeding
* Patient in exclusion period (determined by a previous study or in progress)
* Patient in custody
* Patient under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Comparison of the intra-operative modifications rates | At time of surgery
  Modifications in the surgical planning compared to the plan based on the analysis of standard preoperative images (CT-scan and MRI) and the plan based on the 3D model analysis: changes in surgical resection type (by specifying the surgical act: tumorectomy, segmentectomy, bi-segmentectomy or lobectomy…) or no surgery.

SECONDARY OUTCOMES:
Comparison of tumor(s) location | At time of surgery
  Comparison of tumor(s) location based on 3D model and standard preoperative images analysis.
Comparison of vascular network anatomy | At time of surgery
  Comparison of vascular network anatomy based on 3D model and standard preoperative images analysis.
Choice of surgical plan | At time of surgery
  Surgery done according to a) surgical plan based on standard preoperative images analysis, b) surgical plan based on 3D model analysis or c) alternative approach (by specifying the surgical act: tumorectomy, segmentectomy, bi-segmentectomy or lobectomy….)
Modification of the initial surgical plan, if applicable | At time of surgery
  Description of perioperative events having modified the initial surgical plan.
Comparison of resection merges | At time of surgery
  Comparison of expected resection merges based on standard preoperative images and 3D model analysis and actual resection merge in the operating room.
Comparison of resection volumes | At time of surgery
  Comparison of expected resection volumes based on standard preoperative images and 3D model analysis and actual resection volume in the operating room.
Comparison of surgical merge size | At time of surgery
  Comparison of surgical merge size (mm) based on 3D model and standard preoperative images analysis.
Morbidity | At time of surgery and 3 months after surgery
  Morbidity specific to the procedure.
Mortality | At time of surgery and 3 months after surgery
  Mortality specific to the procedure.
Preoperative images independent analysis | 3 years
  Analysis of preoperative images (CT-scan/MRI and 3D model) by a senior team on one hand, and a junior team (surgeons + radiologists) on the other hand.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Pessaux, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil - Strasbourg
Locations (12):
- France (12):
  - Service de Chirurgie Digestive - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor - Service de Chirurgie Digestive et Hépatobiliaire -, Créteil
  - Service de Chirurgie Digestive et Transplantation - Hôpital Claude Huriez, Lille
  - Service de Chirurgie Digestive et Transplantation Hépatique - Hôpital universitaire de la Croix-Rousse, Lyon
  - Service de Chirurgie Digestive - CH Emile Muller, Mulhouse
  - Chirurgie Viscérale et Digestive - Polyclinique de Gentilly, Nancy
  - Chirurgie Digestive, Hépato-bilio-pancréatique et Transplantation - La Pitié Sâlpêtrière, Paris
  - Service de Chirurgie Digestive - CHU Robert Debré, Reims
  - Service de Chirurgie Digestive Hôpital Charles Nicolle - CHU Rouen, Rouen
  - Institut de Chirurgie Viscérale - Clinique de l'Orangerie, Strasbourg
  - Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil, Strasbourg
  - Centre Hépato-Biliaire - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Background] Gauss T, Merckx P, Brasher C, Kavafyan J, Le Bihan E, Aussilhou B, Belghiti J, Mantz J. Deviation from a preoperative surgical and anaesthetic care plan is associated with increased risk of adverse intraoperative events in major abdominal surgery. Langenbecks Arch Surg. 2013 Feb;398(2):277-85. doi: 10.1007/s00423-012-1028-3. Epub 2012 Nov 13. PMID 23149461
- [Background] Couinaud C. [Errors in the topographic diagnosis of liver diseases]. Ann Chir. 2002 Jun;127(6):418-30. doi: 10.1016/s0003-3944(02)00802-7. French. PMID 12122715
- [Background] Mutter D, Dallemagne B, Bailey Ch, Soler L, Marescaux J. 3D virtual reality and selective vascular control for laparoscopic left hepatic lobectomy. Surg Endosc. 2009 Feb;23(2):432-5. doi: 10.1007/s00464-008-9931-y. Epub 2008 Apr 29. PMID 18443871
- [Background] Mutter D, Soler L, Marescaux J. Recent advances in liver imaging. Expert Rev Gastroenterol Hepatol. 2010 Oct;4(5):613-21. doi: 10.1586/egh.10.57. PMID 20932146